CLINICAL TRIAL: NCT04341792
Title: Predictive Biomarkers of Secondary Aggravation in Covid-19 Suspect Patient Admitted to Emergency Departments During an Epidemic
Brief Title: Predictive Biomarkers of Secondary Aggravation in Covid-19 Suspect Patient
Acronym: BIOCOVU
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_33; 2020-A00906-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Infection Viral; Coronavirus; COVID-19
Keywords: infection viral; biological risk factor; coronavirus; covid-19
MeSH Terms: conditions — Virus Diseases; Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is no predictive tool for patients admitted to the emergency department with a suspicion of Covid-19 that will worsen secondarily and require a heavy lifting.

In a context of saturation of the healthcare system by the pandemic at Covid-19,it is essential to identify specific, accessible prognostic markers via minimally invasive sampling with low risk of infection for personnel caregiver, for optimal allocation of resuscitation resources.

This study proposes to evaluate the biological markers of routine care known to be associated with resuscitation admission in relation to hospitalization on conventional service for the prediction of worsening of patients admitted to the emergencies for Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria for suspicion of Covid-19 in an epidemic period
* Consultation in the emergency departement
* Non-opposition agree

Exclusion Criteria:

* impairment related to another identified cause than Covid-19, in particular a rapid diagnostic test flu-positive
* Severe patient from the outset with transfer to intensive care within 12 hours of admission to the Emergency Department
* No social security coverage (beneficiary or entitled person)
* Poor understanding of French
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population presenting to the emergency department during this pandemic period with symptoms suggestive of Covid-19 infection with no other probable diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Rate of secondary aggravation | an average at 30 days (- 2 days +3 days) of admission to the emergency department
  Secondary aggravation is defined as :
  * a re-hospitalization or
  * aggravation in hospitalization : development or increase in oxygen dependency, hemodynamic failure, and/or respiratory, death

SECONDARY OUTCOMES:
Change of standart biological parameters | Between baseline and an average at 30 days (- 2 days +3 days) of admission to the emergency department
  the number of leukocytes, lymphocytes, neutrophil polynuclear cells, CRP, fibrinogen, and the D-dimers.
Change of Von willebrand factor (vWF) changes over time | Between baseline and an average at 30 days (- 2 days +3 days) of admission to the emergency department
Change of the Factor VIII (FVIII) | Between baseline and an average at 30 days (- 2 days +3 days) of admission to the emergency department
Prevalence of positivity of COVID-19 virus measured by PCR or serology | an average at 30 days (- 2 days +3 days) of admission to the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Garrigue, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU Lille, Lille, France

REFERENCES:
- [Derived] Ledoult E, Guerrier T, Dubucquoi S, Figeac M, Villenet C, Daunou B, Behal H, Pokeerbux MR, Machet T, Koether V, Collet A, Launay D; Lille Covid Research network (LICORNE). Dual role of plasmablasts as immune regulators or amplifiers in COVID-19. Clin Immunol. 2025 Oct 13;281:110609. doi: 10.1016/j.clim.2025.110609. Online ahead of print. PMID 41093046